CLINICAL TRIAL: NCT03328013
Title: Malvacdecision.Net
Brief Title: Impact of HPV Vaccination to Catch up in the Emergence of Lesions of the Cervix
Acronym: HPVAC
Status: Terminated | Type: Observational
Why Stopped: manager's decision
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HPVAC (29BRC17.0086)
Record Dates: First submitted 2017-10-18; First posted 2017-11-01 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: HPV Vaccination; Pap Smear; Cervical Cancer; Catch-up Vaccination
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women aged 25 to 33 years in 2017: Women aged 25 to 33 years in 2017 and having performed an analyzed smear at the Brest University Hospital.
  They are invited to fill out an online questionnaire asking them about :
  * vaccine status against HPV
  * if vaccinated, the name of the vaccine and the number of injection
  * age of first sexual intercourse
  * do they have a gynecological pathology

SUMMARY:
In France, the vaccination coverage observed for HPV vaccination is low for a full-scale regimen, and has been falling since 2010. A high rate of HPV vaccination coverage has a significant epidemiological impact with a reduction in cervical cancer mortality.

There is less data on vaccinated catch-up patients. In 2017, these patients are 25 years of age or older and carry out screening smears.

The aim of this study is to demonstrate whether HPV catch-up vaccination results in a decrease in the abnormal smear rate compared to the rate in unvaccinated patients.

If so, these data will help mobilize doctors to vaccinate patients against HPV, even in catching-up.

DETAILED DESCRIPTION:
In France, the observed vaccination coverage is very low for a complete regimen and has been declining since 2010. This low coverage makes it impossible to benefit from the efficiency observed in the other countries.

Indeed, a high HPV vaccination coverage rate would allow an epidemiologically significant impact with a reduction in cervical cancer mortality. In France, it is estimated that the vaccination of 80% of girls between the ages of 11 and 14 would reduce the incidence of 72% of CIN2 and 54% of CIN3.

Nevertheless, there is less data on patients who have been vaccinated in catch-up. These patients are 25 years of age or older in 2017, and make smears.

The aim of this study is to demonstrate whether HPV catch-up vaccination results in a decrease in the abnormal smear rate compared to the rate in unvaccinated patients.

If our study shows the benefits of catch-up vaccination, these data will help to mobilize doctors to vaccinate girls 15-19 years of age against HPV if they have not been able to benefit between 11 and 14 years as recommended.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged 25 to 33 in 2017
* with a smear analyzed at the Brest University Hospital

Exclusion Criteria:

* men
* age over 33 years or less than 25 years
* patient refusing to participate

Ages: 25 Years to 33 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women, aged 25 to 33 in 2017, with a smear analyzed at the Brest University Hospital, vaccinated or not against HPV
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Nature of smear: normal or not (including ASCUS and AGC) according to their immunization status | Day 1

SECONDARY OUTCOMES:
age of occurrence of lesions according to the year of vaccination | Day 1 (questionnaire completed by patient)
number of injection received | Day 1 (questionnaire completed by patient)
Age of onset of sexual activity | Day 1 (questionnaire completed by patient)
Vaccine received | Day 1 (questionnaire completed by patient)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baudoin A, Sabiani L, Oundjian F, Tabouret E, Agostini A, Courbiere B, Boubli L, Carcopino X. [HPV prophylactic vaccine coverage and factors impacting its practice among students and high school students in Marseilles' area]. J Gynecol Obstet Biol Reprod (Paris). 2015 Feb;44(2):126-35. doi: 10.1016/j.jgyn.2014.02.005. Epub 2014 Apr 2. French. PMID 24703591
- [Background] Doris B, Boyer L, Lavoue V, Riou F, Henno S, Tas P, Sevene L, Leveque J. [Cervical Pap smear in an epidemiologically exposed population: ideas, facts and arguments]. J Gynecol Obstet Biol Reprod (Paris). 2014 Jan;43(1):26-34. doi: 10.1016/j.jgyn.2013.11.012. Epub 2013 Dec 12. French. PMID 24332738
- [Background] Carcopino X, Camus C, Halfon P. [Diagnosis and clinical management of cervical HPV infections]. Presse Med. 2015 Jul-Aug;44(7-8):716-26. doi: 10.1016/j.lpm.2015.02.020. Epub 2015 Jun 9. No abstract available. French. PMID 26067573
- [Background] Wafo E, Ivorra-Deleuze D, Thuillier C, Rouzier R. [Evolution of the awareness of Human Papillomavirus (HPV) in the French population: Results of a telephonic inquiry]. J Gynecol Obstet Biol Reprod (Paris). 2010 Jun;39(4):305-9. doi: 10.1016/j.jgyn.2010.03.007. Epub 2010 Apr 28. French. PMID 20430535
- [Background] Bouvret P, Mougin C, Pretet JL, Meurisse A, Bonnetain F, Fiteni F. [Practices and attitudes regarding HPV vaccination among general practitioners from Besancon]. J Gynecol Obstet Biol Reprod (Paris). 2016 Oct;45(8):972-978. doi: 10.1016/j.jgyn.2015.12.002. Epub 2016 Jan 15. French. PMID 26780841
- [Background] Riethmuller D, Ramanah R, Carcopino X, Leveque J. [The follow up of the women vaccinated against HPV]. J Gynecol Obstet Biol Reprod (Paris). 2013 Oct;42(6):525-33. doi: 10.1016/j.jgyn.2013.03.013. Epub 2013 May 10. French. PMID 23669416
- See also: Related Info — http://www.hcsp.fr/explore.cgi/avisrapportsdomaine?clefr=454
- See also: Related Info — http://www.em-consulte.com/article/943204/vaccination-contre-les-infections-a-papillomavirus
- See also: Related Info — http://www.em-consulte.com/article/989449/epidemiologie-prevention-et-depistage-du-cancer-du
- See also: Related Info — http://www.em-consulte.com/article/798059/article/revision-de-lage-de-vaccination-contre-les-infecti